CLINICAL TRIAL: NCT07134998
Title: A Phase I Study of HRS-6093 Evaluating Safety, Tolerability, and Pharmacokinetics in Participants With Advanced Solid Tumors Harboring KRAS G12D Mutations
Brief Title: Phase I Study of HRS-6093 in Participants With Advanced Solid Tumors Harboring KRAS G12D Mutations
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-6093-101
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-08

CONDITIONS: Advanced KRAS G12D Mutant Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-6093 (Experimental)
  Interventions: Drug: HRS-6093

INTERVENTIONS:
Drug: HRS-6093 — HRS-6093

SUMMARY:
This is an open-label, multi-center phase I clinical study to evaluate HRS-6093 Safety, Tolerability, and Pharmacokinetics in Participants harboring KRAS G12D Mutations with advanced solid tumors. The study consists of dose escalation, dose expansion and efficacy expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood this study and are willing to sign the ICF, with good compliance and cooperation in follow-up;
2. Aged between 18-75 years, with no gender requirement;
3. Participants with histologically/cytologically confirmed advanced solid tumors who have been previously tested or are confirmed by the central laboratory to harbor KRAS G12D mutations; Have failed standard treatment, are intolerant to standard treatment, or have not received standard treatment.
4. ECOG performance status (PS) score of 0 or 1;
5. Life expectancy > 3 months;
6. At least one measurable lesion per RECIST v1.1; A tumor tissue sample must be provided.
7. Adequate organ function

Exclusion Criteria:

1. Toxicity (e.g., gastrointestinal reaction and skin toxicity) from prior anti-tumor treatment has not recovered to Grade ≤ 1 or a level specified in the inclusion/exclusion criteria;
2. Presence of central nervous system (CNS) metastases;
3. Participants with gastrointestinal diseases that affect drug administration/absorption
4. Participants who have undergone major surgery other than diagnosis or biopsy within 28 days before the first dose, or are expected to undergo major surgery during the study period;
5. Presence of serious pulmonary diseases
6. Active tuberculosis or a history of active tuberculosis infection within 48 weeks prior to screening, regardless of whether they have been treated;
7. Active or persistent gastrointestinal bleeding within 6 months prior to screening;
8. History of allogeneic bone marrow or solid organ transplantation;
9. History of deep vein thrombosis or pulmonary embolism within 6 months prior to screening;
10. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring clinical intervention;
11. Positive human immunodeficiency virus (HIV) (HIV1/2 antibodies), active chronic hepatitis B, or active hepatitis C (positive HCV antibody and positive HCV RNA);
12. Known history of hypersensitivity to any component of the drug product to be used in the study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events/serious adverse events (graded as per CTCAE v5.0). | Screening Period to 30 Days After the Last Dose
DLT, | from day1 to day 23; 23 Days
MTD, | from day1 to day 23; 23 Days
RP2D , | 24 months

SECONDARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values | Screening Period to 30 Days After the Last Dose; 24 months
Number of subjects with clinically significant changes in ECOG, vital signs and physical examination. | Screening Period to 30 Days After the Last Dose; 24 months
Number of subjects with changes on ECG. | Screening Period to 30 Days After the Last Dose; 24 months
maximum plasma concentration (Cmax), | Screening Period to Day of the end of treatment/withdrawal. 24 months
time to maximum concentration (Tmax), | Screening Period to Day of the end of treatment/withdrawal. 24 months
area under concentration-time curve from time 0 to the last measurable concentration time point t (AUC0-t), | Screening Period to Day of the end of treatment/withdrawal. 24 months
Area under concentration-time curve from time 0 to infinity (AUC 0-∞), apparent volume of distribution (Vz/F), | Screening Period to Day of the end of treatment/withdrawal. 24 months
elimination half-life (t1/2), and apparent clearance (CL/F); | Screening Period to Day of the end of treatment/withdrawal. 24 months
minimum concentration at steady state (Cmin, ss), | Screening Period to Day of the end of treatment/withdrawal. 24 months
area under the blood concentration-time curve at steady state (AUCss), and accumulation ratio (Rac); | Screening Period to Day of the end of treatment/withdrawal. 24 months
objective response rate (ORR), | Screening Period to PD; 24 months
duration of response (DoR), | Screening Period to PD; 24 months
disease control rate (DCR), | Screening Period to PD; 24 months
progression-free survival (PFS), | Screening Period to PD; 24 months
overall survival (OS). | Screening Period to Day of death of the participant;24months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided